CLINICAL TRIAL: NCT03103555
Title: Treatment of Anti-Interferon-Gamma Autoantibody Associated Acquired Immunodeficiency Syndrome With Bortezomib: Pilot Study
Brief Title: Treatment of Adult-Onset Immunodeficiency With Bortezomib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Treatment AOI with Bortezomib
Record Dates: First submitted 2017-04-01; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Adult-onset Immunodeficiency
Keywords: Anti-interferon gamma autoantibody
MeSH Terms: interventions — Bortezomib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bortezomib and cyclophosphamide (Experimental): Two cycles of bortezomib administered subcutaneously, followed by 4 months of low dose oral cyclophosphamide.
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be subcutaneously administered in 2 treatment cycles with 4 injections of 1.3 mg Bortezomib /m2 body surface per cycle.
  Other Names: Velcade
Drug: Cyclophosphamide — Low dose cyclophosphamide will be given orally for 4 month after completion 2 cycles of bortezomib
  Other Names: Endoxan

SUMMARY:
This is pilot study aimed to investigate the application of proteosome inhibitor, Bortezomib in treatment of patients with neutralizing autoantibody to IFN-γ. The investigators hypothesis is that bortezomib will reduce the antibody level and restore interferon-gamma function, resulting in clinical improvement and should be well-tolerated and safe for use in patients with autoantibody to IFN-γ.

DETAILED DESCRIPTION:
The patients with autoantibody to IFN-γ and past or current history of proven opportunistic infection will receive 2 treatment cycles of bortezomib subcutaneously (4 injections of 1.3 mg Bortezomib /m2 body surface per cycle), followed by low dose oral cyclophosphamide for 4 month after completion treatment with bortezomib.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 60 years
* Positive anti-interferon-gamma autoantibody
* Anti-HIV negative
* Past or current infection with opportunistic infection (OI) such as nontuberculous mycobacteria, proven by culture
* Ability to give written consent, informed written consent
* Negative pregnancy test in premenopausal woman
* Receving antimicrobial for treatment of OI for at least one month.

Exclusion Criteria:

* Pregnancy or lactation
* Absolute neutrophil count <1.5 × 109/ L or platelet count <100× 109/ L or hemoglobin level < 8 g/dL
* Past history of myocardial infarction or heart failure within 6 months before enrollment or prolonged QT interval > 450 msec at screening
* Renal insufficiency (GFR < 30 ml/min)
* Abnormal liver function test (AST> 3 times of UNL)
* Known cancer or receiving other immunosuppressive agent
* Known intolerability to Bortezomib

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Titers of anti-interferon-gamma antibody after treatment with bortezomib | 8 weeks after first dose of bortezomib (after completion 2 cycles of bortezomib)
  Change in titers of anti-interferon-gamma antibody after treatment with
Titers of anti-interferon-gamma antibody after treatment with bortezomib and cyclophosphamide | 1 year after first dose of bortezomib
  Change in titers of anti-interferon-gamma antibody after treatment with bortezomib and cyclophosphamide
Adverse event | 6 months after first dose of bortezomib (after completion 4 months of cyclophosphamide)
  Grade 4 adverse event (probably related)

SECONDARY OUTCOMES:
Disease relapse | 6 month and 1 year after first dose of bortezomib
  Worsening of symptoms and signs

CONTACTS AND LOCATIONS:
Overall Officials: Nasikarn Angkasekwinai, MD., Principal Investigator — Faculty of Mdicine Siriraj Hospital, Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angkasekwinai N, Suputtamongkol Y, Tantibhedhyangkul W, Onlamoon N, Phoompoung P, Pithukpakorn M, Karuphong E, Pusuwan P, Angkasekwinai P. Efficacy of Bortezomib for Treating Anti-Interferon-Gamma Autoantibody-Associated Adult-Onset Immunodeficiency Syndrome. Clin Infect Dis. 2024 Apr 10;78(4):1033-1042. doi: 10.1093/cid/ciad676. PMID 37947190